CLINICAL TRIAL: NCT05139420
Title: Biomarkers of Increased Risk of Developing Metabolic Adaptation to Weight Loss
Brief Title: Risk of Metabolic Adaptation After Weight Loss
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lisa Morselli, MD PhD, Assistant professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO00039217
Record Dates: First submitted 2021-11-18; First posted 2021-12-01 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Weight Loss; Obesity
Keywords: resting metabolic rate; metabolic adaptation
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lifestyle intervention (Experimental): Participants will be enrolled in a weight loss program based on lifestyle changes. They will be given a 6-month subscription to a calorie-reduced meal replacement program that also offers lifestyle coaching.
  Interventions: Other: lifestyle intervention with meal replacement program

INTERVENTIONS:
Other: lifestyle intervention with meal replacement program — participants will be enrolled in a medical weight loss program and will be given a 6 month subscription to a calorie-reduced meal replacement program, in addition to lifestyle advice.

SUMMARY:
This study aims at identifying the neurohormonal biomarkers that characterize individuals at risk of greater metabolic adaptation to weight loss, a disproportionate decline in resting metabolic rate during and after weight loss.

ELIGIBILITY:
Inclusion Criteria:

BMI > or = 30 any ethnicity

Exclusion Criteria:

weight > or = 400 lbs.

diabetes (type 2 or type 1)

hypertension

heart disease

kidney disease

liver disease

active cancer

post solid organ or bone marrow transplant

HIV/AIDS

pregnancy

breastfeeding

current smoker

current recreational drug use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2031-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
change in measured and predicted resting metabolic rate during and after weight loss | 18 months
  resting metabolic rate will be measured by indirect calorimetry every 2 months for 6 months, then every 6 months for an additional 12 month. Predicted resting metabolic rate will be calculated with a mathematical formula at the same time points

SECONDARY OUTCOMES:
change in circulating leptin during and after weight loss | 18 months
  blood will be assayed for this hormone every 2 months for 6 months, then every 6 months for an additional 12 months
change in circulating thyroid hormones during and after weight loss | 18 months
  blood will be assayed for this hormone every 2 months for 6 months, then every 6 months for an additional 12 months
change in circulating GLP-1 during and after weight loss | 18 months
  blood will be assayed for this hormone every 2 months for 6 months, then every 6 months for an additional 12 months
change in circulating PYY during and after weight loss | 18 months
  blood will be assayed for this hormone every 2 months for 6 months, then every 6 months for an additional 12 months
change in circulating AgRP during and after weight loss | 18 months
  blood will be assayed for this hormone every 2 months for 6 months, then every 6 months for an additional 12 months
change in 24h urine catecholamines during and after weight loss | 18 months
  urine will be assayed for these hormones every 2 months for 6 months, then every 6 months for an additional 12 months
change in heart rate variability during and after weight loss | 18 months
  blood will be assayed for this hormone every 2 months for 6 months, then every 6 months for an additional 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa L Morselli, MD PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No